CLINICAL TRIAL: NCT03164369
Title: Accuracy of Real Time 3D Navigation Device to Identify Lumbar Epidural Spacy in Pregnant Patients. A Comparison With Standard Ultrasound.
Brief Title: Real Time 3D Navigation and Traditional US to Identify Epidural Space Depth in Pregnancy
Acronym: Accuro
Status: Completed | Type: Observational
Sponsor: Città di Roma Hospital (Other)
Responsible Party: Principal Investigator, Giorgio Capogna, Head Department of Anesthesia, Città di Roma Hospital
Other Study IDs: 002
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Ultrasound
Keywords: epidural block, ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this double blinded study is to assess the abilities of the SpineNav3DTM technology (Accuro) to identify the lumbar epidural space in parturients using as comparator a standar ultrasound (US) device.

DETAILED DESCRIPTION:
SpineNav3DTM technology facilitates image interpretation of individual 2D lumbar spine scans by automating spinal bone landmark detection and depth measurements and providing a real-time assessment of scan plane orientation in 3D.

Assuming a Type I error rate of 5% (α = 0.05) and a Type II error rate of 20% (β=0.2), a minimum of 76 subjects will be required. All the subjects will have their lumbar area scanned for the measurements of the depth of the epidural space (recorded in cm) by two anesthesiologist, one expert in UD and the other a novice, previously instructed to the use of the Accuro device.

All measurements will be performed either in the sitting or in the supine position at L1/L2, L2/L3 and L3/L4 levels. The expert operator will assess the lumbar spine by using both the devices (standard US and Accuro) while the novice will use only the Accuro.

The primary end-point of the study will be the accuracy of the Accuro to determine the depth of the epidural space using a midline approach using as comparator the measurement obtained with the standard ultrasound device performed by the expert operator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women undergoing antenatal anesthetic consultation

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy single fetus pregnant
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
epidural space depth | day 1
  measurement of the depth of the epidural space

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — Citta di Roma Hospital
Locations (1):
- Citta di Roma Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No